CLINICAL TRIAL: NCT00245258
Title: A Multicenter, Double-Blind Placebo Controlled, Fixed Dose Study With An Open-Label, Flexible Dose Phase To Assess The Efficacy Of Sildenafil Citrate In Providing A Better Sexual Experience Including Quality Of Erections And Satisfaction In Men With Erectile Dysfunction
Brief Title: Study to Evaluate Viagra's Ability to Provide a Better Sexual Experience Through Quality Erections and Satisfaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481239
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate

SUMMARY:
The study objective is to:

1. To evaluate the effect of sildenafil citrate versus placebo on the IIEF_EF Domain at the end of the double-blind phase
2. To assess the relationship between treatment with sildenafil citrate or placebo and responses to the Quality of Erection Questionnaire (QEQ) and Sexual Experience Questionnaire (SEX_Q).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-65.
* Documented clinical diagnosis of erectile dysfunction confirmed by an IIEF-EF Domain score of less than or equal to 25. (If the subject scores greater than 25 on the IIEF-EF Domain, screening procedures should be terminated.)

Exclusion Criteria:

* Subjects who have been treated with more than 6 doses of sildenafil citrate or any other phosphodiesterase type 5 (PDE-5) inhibitor such as vardenafil or tadalafil for erectile dysfunction [Note: subjects should not have taken any PDE-5 inhibitors within 4 weeks prior to the date of screening].

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312
Dates: Start 2005-11; Study Completion 2006-09

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline to Visit 4 (Week 8) in the IIEF Erectile Function (EF) domain score.

SECONDARY OUTCOMES:
The change from baseline to visit 6 (wk 12) in the IIEF-EF domain; the change from baseline to visit 4 (wk 8) and visit 6 (wk 12) in the domains and total score as well as the individual questions of the sexual experience questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Rostov-on-Don
  - Pfizer Investigational Site, Saint Petersburg
- South Korea (2):
  - Pfizer Investigational Site, Pusan
  - Pfizer Investigational Site, Seoul
- Spain (4):
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Seville
- Sweden (4):
  - Pfizer Investigational Site, Karlshamn
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm

REFERENCES:
- [Derived] Cappelleri JC, Tseng LJ, Stecher V, Goldstein I. Enriching the Interpretation of the Erectile Dysfunction Inventory of Treatment Satisfaction: Characterizing Success in Treatment Satisfaction. J Sex Med. 2018 May;15(5):732-740. doi: 10.1016/j.jsxm.2018.03.078. PMID 29699758
- [Derived] Kirby M, Creanga DL, Stecher VJ. Erectile function, erection hardness and tolerability in men treated with sildenafil 100 mg vs. 50 mg for erectile dysfunction. Int J Clin Pract. 2013 Oct;67(10):1034-9. doi: 10.1111/ijcp.12229. PMID 24073975
- [Derived] Claes HIM, Goldstein I, Althof SE, Berner MM, Cappelleri JC, Bushmakin AG, Symonds T, Schnetzler G. Understanding the effects of sildenafil treatment on erection maintenance and erection hardness. J Sex Med. 2010 Jun;7(6):2184-2191. doi: 10.1111/j.1743-6109.2010.01791.x. Epub 2010 Apr 1. PMID 20384942
- [Derived] Loran OB, Stroberg P, Lee SW, Park NC, Kim SW, Tseng LJ, Collins S, Stecher VJ. Sildenafil citrate 100 mg starting dose in men with erectile dysfunction in an international, double-blind, placebo-controlled study: effect on the sexual experience and reducing feelings of anxiety about the next intercourse attempt. J Sex Med. 2009 Oct;6(10):2826-35. doi: 10.1111/j.1743-6109.2009.01428.x. PMID 19817982
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481239&StudyName=Study+to+evaluate+Viagra%27s+ability+to+provide+a+better+sexual+experience+through+quality+erections+and+satisfaction